CLINICAL TRIAL: NCT00134680
Title: Phase II Trial of the Combination of Letrozole 2.5 mg Daily and Trastuzumab 2 mg/kg Weekly in ErbB2 Positive and Estrogen Receptor and/or Progesterone Receptor Positive Metastatic Breast Cancer
Brief Title: Letrozole, Herceptin in Her2neu +, Estrogen Receptor [ER] and/or Progesterone Receptor [PR] Positive, MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1144; 1144-05-6R5 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Breast Cancer
Keywords: estrogen receptor positive; progesterone receptor positive; ErbB2 positive; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole & Trastuzumab (Experimental): Letrozole 2.5 mg tablets daily and Trastuzumab 2 mg/kg by IV weekly
  Interventions: Drug: Letrozole; Drug: Trastuzumab

INTERVENTIONS:
Drug: Letrozole — Letrozole tablets 2.5 mg by mouth daily
  Other Names: Femara
Drug: Trastuzumab — Weekly trastuzumab (4 mg/kg loading dose given by IV over 90 minutes folowed by 2 mg/kg given by IV weekly over 30 minutes, provided the previous dose was well tolerated.
  Other Names: Herceptin

SUMMARY:
The purpose of the study is to investigate the effects (good and bad) that the combination of the drugs letrozole (also called Femara™) and trastuzumab (also called Herceptin®) has on breast cancer. The United States (US) Food and Drug Administration has approved both letrozole and Herceptin for the treatment of advanced breast cancer. Doctors hope that the combination will work better than either drug alone.

DETAILED DESCRIPTION:
Since ER function is regulated by peptide growth factor signaling, the phenotype of ER positive tumors may be influenced by the expression of growth factors and growth factor receptors. A potential interaction between ErbB2 (HER2/neu) expression and the success of endocrine therapy has been examined. ErbB2 expression was shown to correlate with resistance to hormone therapy.

An inverse relationship between endocrine therapy responsiveness and ErbB2 expression has not been observed in all studies. This may be due to discordant ER status between the primary tumor and metastatic sites. ER status can be discordant in approximately 20% of cases, with a tendency for metastatic disease to become ER negative with time. Data concerning ErbB2 is more limited, but there may be similar lack of concordance between primary tumor and metastases.

Inhibition of ErbB2 signaling may slow the development of resistance to estrogen deprivation therapy by inhibiting a pathway that promotes estrogen independent growth. The ErbB2 signal transduction pathway bypasses the requirement for estrogen for breast epithelial cell growth. When ErbB2 is activated in ER positive breast cancer cells in vitro, ER becomes phosphorylated and capable of stimulating transcription without estrogen. Chronic activation with heregulin, a ligand for the ErbB family of receptors, leads to ER down-regulation and the acquisition of an ER negative phenotype.

Estrogen deprivation therapy with selective aromatase inhibitors (SAIs) has become the standard of care for postmenopausal women with tamoxifen-resistant advanced breast cancer. About 1/3 of patients benefit from this therapy. There is interest in treating endocrine therapy refractory breast cancer with the recombinant DNA-derived humanized monoclonal antibody trastuzumab. When given alone, trastuzumab has an endocrine therapy-like risk benefit ratio. Trastuzumab targets ErbB2 (HER2/neu). Some breast cancers may coexpress ER and ErbB2.

Letrozole (Femara™) is a highly selective oral non-steroidal aromatase inhibitor. According to in vitro data, letrozole is 170-fold more potent in inhibiting aromatase than aminoglutethimide (AG) and 19-fold more active than anastrozole. Letrozole effectively inhibits intratumoral aromatase according to in vitro and in vivo data. It is indicated for the treatment of advanced breast carcinoma in post-menopausal women who have failed prior anti-estrogen therapy. Final FDA approval was granted in 1997. In two randomized phase IIb/III studies in patients previously treated with an antiestrogen, 19.5% and 23.6% of patients achieved an objective response with letrozole 2.5 mg/day compared with 12.4% receiving AG and 16.4% of patients receiving megace. Median overall survival was increased in the letrozole 2.5 mg/day group by 8 months compared to AG and by 3 months compared to megace. The lower 0.5 mg/day dose of letrozole was associated with poorer response rates and overall survival in both studies.

Trastuzumab (Herceptin®) was approved in 1998. A trial of trastuzumab as a single agent for first line treatment of advanced disease has been reported. Response rate in the first 62 patients was 24%.

The primary objective of this trial is to determine the proportion of patients with ER and/or PR positive, ErbB2 positive tamoxifen resistant metastatic breast cancer who achieve complete remission or partial remission or no significant change in lesion size for > 24 weeks from a combination of letrozole and trastuzumab. The study will also determine duration of response and median time to progression, evaluate toxicity, generate a tumor and serum bank, and analyze ErbB2 expression on circulating malignant cells during treatment.

The study will enroll 35 patients

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal.
* If premenopausal at diagnosis, eligible if undergoes treatment with luteinising hormone-releasing hormone (LHRH) agonist or surgical ovarian ablation before initiating treatment (tx).
* Tumor cell expression of ER and/or PR and ErbB2. Expression can be ascertained on either primary or metastatic site.
* Patient may have received adjuvant and/or neoadjuvant chemotherapy.
* Patient who received adjuvant/neoadjuvant chemotherapy, tx. must have been discontinued for 4 weeks and patient must have recovered from all acute toxicities, except alopecia.
* Prior radiotherapy is permitted as long as it was planned before start of study medication and is completed within 3 weeks of starting trial medication.
* Prior megestrol acetate or raloxifene therapy is permitted, but must be stopped prior to trial entry.
* Prior tamoxifen therapy.
* At least one bidimensionally measurable lesion.
* ECOG performance status 0-2.
* Patient should have life expectancy of 6 months.
* Patient must have adequate hematologic function: absolute neutrophil count (ANC) 1000/mm3; platelets 75,000/mm3.
* Patient must have adequate renal and liver function, defined as: serum creatinine less than or equal to 1.5 times the upper limit of normal; serum bilirubin less than or equal to 1.5 times the upper limit of normal (three times the upper limit of normal for patients with hereditary benign hyperbilirubinaemia); transaminases (ALT, AST) less than or equal to 2.5 times the upper limit of normal in patients without liver metastasis, or less than or equal to 5 times the upper limit of normal in patients with liver metastasis.
* Ejection fractions by multiple-gated acquisition (MUGA) scan or echocardiogram greater than 50%
* Patient must give written informed consent prior to initiation of any invasive study-related procedures that would otherwise not be performed, and must be able to comply with scheduled visits and evaluations.
* Treatment with bisphosphonates during the trial is permitted.

Exclusion Criteria:

* Prior exposure to any aromatase inhibitor (aminoglutethimide, formestane anastrozole, letrozole or exemestane) for more than 28 days. Patients that have already started on aromatase inhibitors (AIs) will be eligible for the protocol if they meet all other eligibility requirements and receive loading dose of trastuzumab not more than 28 days after starting AI therapy. Patients who initially received anastrozole or exemestane will be switched to letrozole.
* Prior treatment with trastuzumab
* Prior anthracycline exposure in adjuvant setting > 360 mg/m2.
* Patients with central nervous system (CNS) involvement with metastatic breast cancer or life threatening lymphangitic or large volume lung or liver disease.
* Patient's only qualifying lesions have been previously irradiated or are scheduled for irradiation following study entry.
* Severe or uncontrolled concomitant disease from other causes.
* More than 1 prior course of chemotherapy for metastatic disease. If patient has received one course of palliative chemotherapy, acute toxicities must have resolved and patient must be experiencing progressive disease at time of enrollment.
* ECOG performance status 3 or 4.
* Patient has previous malignancies other than breast cancer except:

  * adequately treated in situ carcinoma of cervix;
  * localized basal or squamous cell carcinoma of skin; or
  * any previous malignancy treated with curative intent with recurrence risk of less than 30%.
* Patient is unable to understand informed consent or is unlikely to be compliant with protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2000-01; Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients with ER and/or PR positive, ErbB2 positive tamoxifen resistant metastatic breast cancer who achieve complete remission (CR)
or partial remission (PR)
or no significant change in lesion size for greater than 24 weeks

SECONDARY OUTCOMES:
To determine duration of response and median time to progression with letrozole plus trastuzumab treatment
To evaluate the clinical adverse experience during treatment with letrozole plus trastuzumab treatment
To generate a tumor and serum bank from patients receiving combination trastuzumab and letrozole treatment
To analyze ErbB2 expression on circulating malignant cells during treatment with letrozole and trastuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Marcom, MD, Principal Investigator — Duke University; Matthew J Ellis, MB, PhD, Study Director — Washington University School of Medicine
Locations (4):
- United States (4):
  - Lombardi Cancer Institute, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center, Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Result] Marcom PK, Isaacs C, Harris L, Wong ZW, Kommarreddy A, Novielli N, Mann G, Tao Y, Ellis MJ. The combination of letrozole and trastuzumab as first or second-line biological therapy produces durable responses in a subset of HER2 positive and ER positive advanced breast cancers. Breast Cancer Res Treat. 2007 Mar;102(1):43-9. doi: 10.1007/s10549-006-9307-8. Epub 2006 Aug 8. PMID 16897431